CLINICAL TRIAL: NCT06048198
Title: Incidence and Predictors of Delirium in the Trauma Intensive Care Unit：Prospective Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202307121RINC
Record Dates: First submitted 2023-09-10; First posted 2023-09-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Delirium, Risk Factor
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background Delirium is an acute neuropsychiatric syndrome, and its causes remain complex and not fully comprehended. Patients in trauma intensive care units are at high risk for delirium and are greatly affected by its adverse outcomes. As there are currently no effective pharmacological treatments or approaches for delirium, it is crucial to focus on identifying the risk factors for delirium and implementing early prevention strategies.

Objective Analyzing the incidence and risk factors of delirium in trauma intensive care unit patients.

Method This study is a prospective research that focuses on all patients in the trauma intensive care unit of a medical center. Data collection will be conducted through questionnaires and electronic medical records. A total of 200 participants will be conveniently selected for the study. Upon admission to the intensive care unit, each patient will complete a basic information questionnaire, and their medical records will be collected daily until they are discharged from the intensive care unit. The study incorporates various assessment scales including Intensive Care Delirium Screening Checklist (ICDSC), Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), Acute Physiology and Chronic Health Evaluation II (APACHE-II), Injury Severity Score (ISS), and Malnutrition Universal Screening Tool (MUST). Statistical analysis will be done by using IBM SPSS 24.0 for Windows. Descriptive statistics including mean, standard deviation, and percentages will be used to present demographic information. Logistic regression analysis will be applied to identify the key predictive factors for delirium risk.

Expected outcome and clinical application This study anticipates that the non-modifiable risk factors for trauma intensive care unit patients include age, substance use, chronic diseases, traumatic brain injury, prior surgery, frailty, APACHE II score, ISS, and ASA anesthesia classification. The modifiable risk factors include malnutrition, polypharmacy, electrolyte deficiency, metabolic acidosis, pain, mechanical ventilation, physical restraints, total surgical duration, intraoperative blood loss, and low hemoglobin. By understanding these risk factors, high-risk patients can be identified and preventive measures can be implemented to reduce the occurrence of delirium. Furthermore, addressing modifiable risk factors can help in reducing the risk or severity of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to trauma intensive care unit.
* Age ≥18.
* Patients who belongs to surgical or trauma subject.

Exclusion Criteria:

* Patients who stay in trauma ICU less than 24hrs.
* Patients who can not communicate with Chinese or Taiwanese.
* Patients who was diagnosed dementia.
* Patients who was evaluated -4 or -5 on Richmond Agitation-Sedation Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who admitted to trauma intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Delirium incidence | once per day
  The incidence of delirium in the trauma ICU.
Predictors of delirium | once per 2-days
  The risk factors of delirium in the trauma ICU.(Age, APACHE II, ISS, MUST, 5-mFI, blood exam data...)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, 臺灣, Taiwan

IPD SHARING:
Plan to Share IPD: No